CLINICAL TRIAL: NCT05962047
Title: Use of Augmented Reality for Restricted and Repetitive Behavior and Executive Function of Children With Autism Spectrum Disorder
Brief Title: Augmented Reality for Behavior and Executive Function of Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F723 - Project A
Record Dates: First submitted 2023-06-26; First posted 2023-07-27 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Autism Spectrum Disorder
Keywords: Augmented Reality; Behaviour; Executive function
MeSH Terms: conditions — Autism Spectrum Disorder; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcome assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Augmented Reality games
  Interventions: Other: Games of WonderTree Augmented Reality
- Group 2 (Active Comparator): Traditional therapy
  Interventions: Other: Traditional therapy

INTERVENTIONS:
Other: Games of WonderTree Augmented Reality — Participants of group 1 (experimental group) will augmented reality based interventions comprising of games of Wonder Tree
  Arms: Group 1
Other: Traditional therapy — Traditional therapy based on play activities utilizing blocks, colors, Velcro-based toys.
  Arms: Group 2

SUMMARY:
The aim of the study is to determine the effects of usage of augmented reality for Restricted and repetitive behavior and executive function of children with autism spectrum disorder

DETAILED DESCRIPTION:
Augmented Reality allows children to see a representation of imaginary content and pretend play overlaid on the real-world environment. Today, technology can be a safe and motivating way of engaging children with autism in social interaction activities. Current research in therapeutic technology for autism is aimed toward improving behavior and psychomotor activities that impact social communication. The aim of this research project is to help teachers, parents, practitioners, and researchers to understand the unique strengths of their children with autism along with technology based educational and therapeutic activities for home and classroom.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with autism spectrum disorder in the age range of 5-12 years at verbal imitation and 1-step command following.

Exclusion Criteria:

* Sensory issues and patients on medication

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Developmental Behaviour Checklist (DBC) | After 8 weeks
  The Developmental Behaviour Checklist (DBC) can be used for the assessment of behavioural and emotional problems of children and adolescents with development and intellectual disabilities. It is a questionnaire completed by parents or other primary carers, or teachers and reports problems over a six month period

SECONDARY OUTCOMES:
Repetitive Behaviors Scale-Revised (RBS-R) | After 8 weeks
  The RBS-R is a 44-item self-report questionnaire that is used to measure the breadth of repetitive behavior in children, adolescents, and adults with Autism Spectrum disorders.
The flexibility Scale | After 8 weeks
  Cognitive flexibility is the ability to switch between different thoughts and actions. It is considered part of executive functions, which are the general mental functions that help us to coordinate thought and action. The tool has a four point ordinal likert scale scoring for each item. Higher scores (after reverse scoring) mean greater endorsement of problems / characteristics.
Digital span memory test | After 8 weeks
  Digital span test will be used to determine working memory. It is a working memory test that is used in many cognitive and neuroscience research labs. Th patient is instructed to repeat the sequence of numbers shown during the test. To make it more interesting, gradually increase the Span, which starts out at 8, and change to Fast test speed. The Digit Span score is the length of the longest correctly repeated sequence
The Stroop test | After 8 weeks
  The Stroop test also known as the color-word naming test, will be used for cognitive inhibition. It is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference.
  The basic Stroop scores (time taken in seconds for each of the three cards) will be entered. Subjects (S's) basic score on each card is the total time (in seconds) to utter the 100 names.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Child Development Center - Riphah International University, Islamabad, AL, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berenguer C, Baixauli I, Gomez S, Andres MEP, De Stasio S. Exploring the Impact of Augmented Reality in Children and Adolescents with Autism Spectrum Disorder: A Systematic Review. Int J Environ Res Public Health. 2020 Aug 24;17(17):6143. doi: 10.3390/ijerph17176143. PMID 32847074
- [Background] Dechsling A, Orm S, Kalandadze T, Sutterlin S, Oien RA, Shic F, Nordahl-Hansen A. Virtual and Augmented Reality in Social Skills Interventions for Individuals with Autism Spectrum Disorder: A Scoping Review. J Autism Dev Disord. 2022 Nov;52(11):4692-4707. doi: 10.1007/s10803-021-05338-5. Epub 2021 Nov 16. PMID 34783991